CLINICAL TRIAL: NCT01015716
Title: Physical Exercise, Dietary Counseling and Cognitive Behavioral Training as a Combined Life-style Intervention to Reduce Weight and Increase Workability in Health Care Workers
Brief Title: Physical Exercise, Dietary Counseling and Cognitive Behavioral Training as a Combined Intervention to Reduce Weight and Increase Workability in Health Care Workers
Acronym: FINALE-Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Working Environment Research Foundation (Unknown); The Ministry of Culture Committee on Sports Research, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FINALE-Health
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Overweight; Physical Capacity; Musculoskeletal Diseases; Work Ability; Sick-leave
Keywords: Weight loss; Physical activity; Cognitive Behavioral Training
MeSH Terms: conditions — Overweight; Musculoskeletal Diseases; Weight Loss; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control-group (Active Comparator): Invitation to attend a monthly seminar of 2 hour duration on a wide range of health related topics
  Interventions: Behavioral: Control-group
- Intervention-group (Experimental): Physical exercise, dietary counseling and cognitive behavioral training as a combined intervention
  Interventions: Behavioral: Intervention-group

INTERVENTIONS:
Behavioral: Intervention-group — Physical exercise, dietary counseling and cognitive behavioral training as a combined intervention
  Arms: Intervention-group
Behavioral: Control-group — Invitation to attend a monthly seminar of 2 hour duration on a wide range of health related topics
  Arms: Control-group

SUMMARY:
The purpose of this study is to evaluate whether a 1 year worksite based life-style intervention can reduce body weight and increase physical capacity and subsequently reduce musculoskeletal disorders and increase workability in overweight health care workers.

DETAILED DESCRIPTION:
Health care workers have a high rate of musculoskeletal disorders and sick leave and a poor workability and physical fitness. Most studies have focused on increasing physical fitness in order to increase workability and to reduce musculoskeletal disorders and sick leave. Studies however also show that many health care workers are obese and obesity has been linked to poor workability.

Limited research is available on the effect of reducing body-weight in this group in order to increase workability and to decrease musculoskeletal disorders and sick leave.

This study introduces a combined worksite based lifestyle intervention consisting of physical exercise, dietary counseling and cognitive behavioral training aimed at reducing weight in health care workers.

On specific worksites, health care workers are cluster randomized to either intervention or control group.

Effects on physical capacity, body composition, musculoskeletal disorders, workability and sick leave are evaluated before and after a 1 year intervention period

ELIGIBILITY:
Inclusion Criteria:

* Overweight Health care workers, working more than 15 hours pr week

Exclusion Criteria:

* Pregnancy, angina pectoris and life-threatening diseases according to safty regulations for physical evaluation methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
weight loss | 3 months
Weight loss | 1 year

SECONDARY OUTCOMES:
Muscle strength | 3 months
Aerobic capacity | 3 months
Health Check | 1 year
Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette R. Christensen, M.Sc. PT, Principal Investigator — Department of Sport Science
Locations (1):
- Department of Sport Science, Aarhus, Denmark

REFERENCES:
- [Derived] Christensen JR, Pajevic M, Ilvig PM, Sogaard K, Jessen-Winge C. Why people engage in a weight loss intervention at their workplace - a stratified case study. BMC Public Health. 2019 Jan 7;19(1):20. doi: 10.1186/s12889-018-6346-0. PMID 30612549
- [Derived] Christensen JR, Kongstad MB, Sjogaard G, Sogaard K. Sickness Presenteeism Among Health Care Workers and the Effect of BMI, Cardiorespiratory Fitness, and Muscle Strength. J Occup Environ Med. 2015 Dec;57(12):e146-52. doi: 10.1097/JOM.0000000000000576. PMID 26641838
- [Derived] Christensen JR, Overgaard K, Carneiro IG, Holtermann A, Sogaard K. Weight loss among female health care workers--a 1-year workplace based randomized controlled trial in the FINALE-health study. BMC Public Health. 2012 Aug 8;12:625. doi: 10.1186/1471-2458-12-625. PMID 22871173
- [Derived] Christensen JR, Faber A, Ekner D, Overgaard K, Holtermann A, Sogaard K. Diet, physical exercise and cognitive behavioral training as a combined workplace based intervention to reduce body weight and increase physical capacity in health care workers - a randomized controlled trial. BMC Public Health. 2011 Aug 27;11:671. doi: 10.1186/1471-2458-11-671. PMID 21871113
- [Derived] Holtermann A, Jorgensen MB, Gram B, Christensen JR, Faber A, Overgaard K, Ektor-Andersen J, Mortensen OS, Sjogaard G, Sogaard K. Worksite interventions for preventing physical deterioration among employees in job-groups with high physical work demands: background, design and conceptual model of FINALE. BMC Public Health. 2010 Mar 9;10:120. doi: 10.1186/1471-2458-10-120. PMID 20214807